CLINICAL TRIAL: NCT04419038
Title: Evaluation of Conjunctival Autografting Augmented With Mitomycin-C Application Versus Ologen Implantation in Surgical Treatment of Recurrent Pterygium
Brief Title: Evaluation of Conjunctival Autografting With MMC Application Versus Ologen Implantation of Recurrent Pterygium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amin Faisal Ellakwa, clinical professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81046
Record Dates: First submitted 2020-05-14; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Recurrent Pterygium of Eye
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conjunctival autografting with MMC (Active Comparator): Group A included 32 eyes of 32 patients who underwent conjunctival autografting augmented with topical application of Mitomycin C (0.2 mg/mL).
  Interventions: Procedure: conjunctival autografting augmented with topical application of Mitomycin C; Procedure: conjunctival autografting augmented with Ologen implantation
- conjunctival autografting augmented with Ologen implantation (Active Comparator): Group B included 31 eyes of 31 who underwent conjunctival autografting augmented with Ologen implantation.
  Interventions: Procedure: conjunctival autografting augmented with topical application of Mitomycin C; Procedure: conjunctival autografting augmented with Ologen implantation

INTERVENTIONS:
Procedure: conjunctival autografting augmented with topical application of Mitomycin C — Group A included 32 eyes of 32 patients who underwent conjunctival autografting augmented with topical application of Mitomycin C (0.2 mg/mL).
Procedure: conjunctival autografting augmented with Ologen implantation — Group B included 31 eyes of 31 who underwent conjunctival autografting augmented with Ologen implantation.

SUMMARY:
Ologen implantation with conjunctival autografting shows promising results in surgical management of recurrent pterygium comparable to MMC application with conjunctival autografting with mild non vision threatening postoperative complications.

DETAILED DESCRIPTION:
Patients were randomly enrolled into two groups. Group A included 32 eyes of 32 patients who underwent conjunctival autografting augmented with topical application of Mitomycin C (0.2 mg/mL). Group B included 31 eyes of 31 who underwent conjunctival autografting augmented with Ologen implantation.

All patients had a recurrent nasal pterygium after one surgical session for removal of the primary one. Any patient with primary nasal pterygium, or patients with recurrent pterygium who had more than one session for surgical removal were excluded. As well, patients with cicatrizing conjunctival disease or previous conjunctival surgery were excluded from the study.

A comprehensive ophthalmic examination, including best-corrected visual acuity testing, slit-lamp examination, Goldmann applanation tonometry, fundus examination, and examination of ocular motility, was carried out for all patients. According to their corneal extent, pterygia were classified into 3 grades:

Grade 1: Fibrovascular proliferations extend up to one quarter of the corneal diameter.

Grade 2: Fibrovascular proliferations extend up to the center of the cornea. Grade 3: Fibrovascular proliferations extend beyond the visual axis.

Consents were taken from all patients and research was approved by the institutional review board. All measures were in accordance with the tenets of the Declaration of Helsinki.

As for group A, 0.2 mg/mL MMC was prepared by reconstituting 2 mg vial of Mitomycin with 10 mL sterile water for injection. When using Mitomycin 10 mg vial, the same concentration was achieved by reconstituting the 10 mg vial 10 mL sterile water for injection. Then 1 ml of the prepared solution was diluted with 4 ml of saline to achieve 0.2 mg/mL (0.02% solution). This solution is stable for 2 weeks under refrigeration, and 24 hours at room temperature (59° to 86°F).

As for group B, 1×2 or 2×2 square millimeter porous collagen matrix was used for each patient

ELIGIBILITY:
Inclusion Criteria:

recurrent nasal pterygium after one surgical session for removal of the primary one

Exclusion Criteria:

* primary nasal pterygium,
* recurrent pterygium with more than one session for surgical removal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
32 eyes with Topical application of Mitomycin C in concentration of (0.2 mg/mL). | "through study completion, an average of 1 year".
  As for group A, 0.2 mg/mL MMC was prepared by reconstituting 2 mg vial of Mitomycin with 10 mL sterile water for injection. When using Mitomycin 10 mg vial, the same concentration was achieved by reconstituting the 10 mg vial 10 mL sterile water for injection. Then 1 ml of the prepared solution was diluted with 4 ml of saline to achieve 0.2 mg/mL (0.02% solution).
31 eyes with ologen implantation(6 mm in diameter and 2 mm thick.) was used for each patient. | "through study completion, an average of 1 year".
  In group B; Ologen was applied under the graft tissue once it is secured in place (half the vial is used for every patient)

REFERENCES:
- [Derived] Wagdy FM, Farahat HG, Ellakwa AF, Mandour SS. Evaluation of Conjunctival Autografting Augmented with Mitomycin C Application versus Ologen Implantation in the Surgical Treatment of Recurrent Pterygium. J Ophthalmol. 2021 Jan 12;2021:8820926. doi: 10.1155/2021/8820926. eCollection 2021. PMID 33505715